CLINICAL TRIAL: NCT06965023
Title: Microplastics and Nanoplastics (MNPs) in Patients With ST-elevation Myocardial Infarction (STEMI)
Acronym: STEMI-Plastics
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera "Sant'Andrea" (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Morgagni Pierantoni Hospital (Other); Azienda Ospedaliera Sant'Anna e San Sebastiano (Other); University Hospital, Catania (Other); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); Niguarda Hospital (Other); Azienda Ospedaliera Universitaria Ferrara (Unknown)
Responsible Party: Principal Investigator, Emanuele Barbato, Full Professor, Azienda Ospedaliera "Sant'Andrea"
Other Study IDs: 0379/2025
Record Dates: First submitted 2025-04-23; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: ST-elevation Myocardial Infarction (STEMI); Microplastics; Nanoplastics; Pollution Exposure
Keywords: STEMI; Microplastics; Nanoplastics; Inflammation; OCT; Plaque composition; cardiac magnetic resonance; Pollution; Exposome; Infarct Size; Coronary Microvascular Dysfunction; IMR; MRR
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI patients with presence of micro- and nano-plastics (MNPs).: Consecutive patients with ST-elevation myocardial infarction (STEMI) undergoing urgent invasive coronary angiography with evidence of acute thrombotic coronary occlusion/sub-occlusion and clinical indication to thromboaspiration with the presence of micro- and nano-plastics (MNPs).
- STEMI patients without presence of micro- and nano-plastics (MNPs): Consecutive patients with ST-elevation myocardial infarction (STEMI) undergoing urgent invasive coronary angiography with evidence of acute thrombotic coronary occlusion/sub-occlusion and clinical indication to thromboaspiration without the presence of micro- and nano-plastics (MNPs).

SUMMARY:
Air pollution and microplastics pose major public health threats. Emerging data have shown that micro- and nanoplastics (MNPs) are ubiquitous environmental pollutants accumulating in human tissues, triggering inflammation and prothrombotic state. This study will investigate the presence and burden of MNPs within coronary thrombi/thromboaspirate of patients presenting with ST segment elevation acute myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention and their association with cardiac damage, plaque vulnerability, microvascular obstruction, and cardiovascular events. Plaque vulnerability will be explored by optical coherence tomography, while microvascular obstruction will be assessed by bolus thermodilution and cardiac magnetic resonance. Participants will be followed up for 1-year to evaluate whether the presence and the burden of MNPs will be associated with a higher incidence of the cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

All the following inclusion criteria should be fulfilled:

1. Age > 18 years old;
2. STEMI undergoing urgent invasive coronary angiography;
3. Acute thrombotic coronary occlusion/sub-occlusion (TIMI 0/1);
4. Clinical indication to thromboaspiration;
5. Able to give informed consent.

Exclusion Criteria:

1. Contraindications to percutaneous coronary intervention;
2. Hemodynamic instability or cardiogenic shock;
3. End-stage chronic kidney disease;
4. Life expectancy < 1 year due to non-cardiac pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with ST-elevation myocardial infarction (STEMI) undergoing urgent invasive coronary angiography with evidence of acute thrombotic coronary occlusion/sub-occlusion and clinical indication to thromboaspiration will be considered eligible for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate in STEMI patients. | From enrollment until the date of hospital discharge, assessed up to 7 days
  To assess the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate of patients experiencing an ST-elevation myocardial infarction.
Correlation of micro- and nanoplastics (MNPs) in coronary thromboaspirate in STEMI patients with inflammatory and cardiac damage biomarkers. | From enrollment until the date of hospital discharge, assessed up to 7 days
  To assess the correlation between the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate of patients experiencing an ST-elevation myocardial infarction with inflammatory, oxidative stress, and cardiac damage biomarkers of peripheral and coronary blood samples.

SECONDARY OUTCOMES:
Burden of micro- and nanoplastics (MNPs) in culprit vs. non-culprit vessels. | From enrollment until the date of hospital discharge, assessed up to 7 days
  To assess the difference in the burden of micro- and nanoplastics (MNPs) between the culprit coronary artery and the contralateral coronary artery.
Age- and sex- related differences in the burden of micro- and nanoplastics (MNPs). | From enrollment until hospital discharge (up to 7 days from enrollment)
  To evaluate the variation in the burden of micro- and nanoplastics (MNPs) based on sex and across different age groups.
Burden of micro- and nanoplastics (MNPs) in STEMI patients across different geographic regions. | From enrollment until hospital discharge (up to 7 days from enrollment).
  To evaluate the variation in the burden of micro- and nanoplastics (MNPs) across different geographic regions.
Association of burden of micro- and nanoplastics (MNPs) with air pollution. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) with air pollution across different geographic regions.
Differences in the burden of micro- and nanoplastics (MNPs) across biological samples. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To assess differences in the burden of micro- and nanoplastics (MNPs) across venous blood, arterial blood, and urine samples.
Micro- and nanoplastics (MNPs) in diabetic vs. non-diabetic patients. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To assess the difference in the burden of micro- and nanoplastics (MNPs) between diabetic and non-diabetic patients.
Micro- and nanoplastics (MNPs) in patients with and without chronic kidney disease. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To assess the difference in the burden of micro- and nanoplastics (MNPs) between patients with and without chronic kidney disease.
Micro- and nanoplastics (MNPs) clearance in patients with and without chronic kidney disease. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To evaluate the clearance of micro- and nanoplastics (MNPs) assessed through plasma and urine concentration measurements of MNPs in patients with and without chronic kidney disease.
  The clearance of MNPs will be quantified by comparing concentrations of identified micro- and nanoplastics in plasma and urine samples collected at the defined time points. Clearance will be estimated based on MNP plasma decay curves and cumulative urinary excretion.
Variation in the burden of micro- and nanoplastics (MNPs) between baseline and follow-up. | From enrollment to follow-up.
  To evaluate the variation in the burden of micro- and nanoplastics (MNPs) between baseline and follow-up in venous blood samples.
Association of the burden of micro- and nanoplastics (MNPs) with coronary reperfusion. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) with the success of coronary reperfusion as assessed by TIMI flow and MBG at invasive coronary angiography.
Association of the burden of micro- and nanoplastics (MNPs) with plaque composition as assessed by optical coherence tomography (OCT). | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with plaque composition as assessed by intravascular imaging (optical coherence tomography - OCT).
Association of the burden of micro- and nanoplastics (MNPs) with microvascular dysfunction/obstruction post PCI as assessed by invasive bolus thermodilution. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) with microvascular dysfunction/obstruction post percutaneous coronary intervention as assessed by invasive bolus thermodilution.
Association of the burden of micro- and nanoplastics (MNPs) with infarct size, myocardial area at risk, microvascular obstruction, and intramyocardial hemorrhage at cardiac magnetic resonance (CMR). | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) with infarct size, myocardial area at risk, microvascular obstruction, and intramyocardial hemorrhage as assessed by cardiac magnetic resonance (CMR).
Association of the burden of micro- and nanoplastics (MNPs) with peak Troponin. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with the peak value of high-sensitivity troponin (hs-Tn).
Association of the burden of micro- and nanoplastics (MNPs) with left ventricular ejection fraction and wall motion score index at echocardiography. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with left ventricular ejection fraction and wall motion score index as assessed by echocardiography at hospital admission and discharge.
Association of the burden of micro- and nanoplastics (MNPs) with in-hospital arrhythmic burden. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with the in-hospital arrhythmic burden.
Association of the burden of micro- and nanoplastics (MNPs) with in-hospital cardiovascular death. | From enrollment until hospital discharge (up to 7 days from enrollment)
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with in-hospital cardiovascular death.
Association of the burden of micro- and nanoplastics (MNPs) with left ventricular recovery at 3 months follow-up. | From enrollment to 3-month follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with left ventricular recovery at 3-month follow-up as assessed by echocardiography.
Association of the burden of micro- and nanoplastics (MNPs) with recurrence angina at 3-month follow-up. | From enrollment to 3-month follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with the recurrence of angina at 3-month follow-up.
Association of the burden of micro- and nanoplastics (MNPs) with all-cause death at 1-year follow-up. | From enrollment to 1 year follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with all-cause death at 1-year follow-up.
Association of the burden of micro- and nanoplastics (MNPs) with cardiovascular death at 1-year follow-up. | From enrollment to 1 year follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with cardiovascular death at 1-year follow-up.
Association of the burden of micro- and nanoplastics (MNPs) with hospitalization for heart failure at 1-year follow-up. | From enrollment to 1 year follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with hospitalization for heart failure at 1-year follow-up.
Association of the burden of micro- and nanoplastics (MNPs) with the recurrence of myocardial infarction at 1-year follow-up. | From enrollment to 1 year follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with the recurrence of myocardial infarction at 1-year follow-up.
Association of the burden of micro- and nanoplastics (MNPs) with target vessel failure at 1-year follow-up. | From enrollment to 1 year follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with target vessel failure at 1-year follow-up.
Association of the burden of micro- and nanoplastics (MNPs) with major adverse cardiovascular events (MACE) at 1-year follow-up. | From enrollment to 1 year follow-up.
  To correlate the burden of micro- and nanoplastics (MNPs) in coronary thromboaspirate with major adverse cardiovascular events (MACE) at 1-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Paolisso, MD, PhD, Study Chair — Sant'Andrea University Hospital; Marta Belmonte, MD, Study Chair — Sant'Andrea University Hospital
Locations (10):
- Italy (10):
  - Sant'Andrea University Hospital, Roma, Rome
  - Department of Environmental Biological and Pharmaceutical Sciences and Technologies, University of Campania "Luigi Vanvitelli, Caserta
  - Division of Cardiology, A.O.R.N. "Sant'Anna e San Sebastiano", Caserta, Italy., Caserta
  - Cardiovascular Department, A.O.U. Policlinico "G. Rodolico - San Marco", University of Catania, Catania, Italy., Catania
  - Azienda Ospedaliero Universitaria di Ferrara, Cona, Italy, Ferrara
  - Cardiovascular Division, Morgagni-Pierantoni University Hospital, Forlì, Italy., Forlì
  - Interventional Cardiology Unit, De Gasperis Cardio Center, Niguarda Hospital, Milan, Italy., Milan
  - Department of Advanced Medical and Surgical Sciences, University of Campania-Luigi Vanvitelli, Naples, Italy., Naples
  - Division of Cardiology, Cardiovascular and Thoracic Department, Città della Salute e della Scienza, Turin, Italy., Turin
  - Azienda Ospedaliera Integrata Verona, Italy, Verona

REFERENCES:
- [Background] Liu S, Wang C, Yang Y, Du Z, Li L, Zhang M, Ni S, Yue Z, Yang K, Wang Y, Li X, Yang Y, Qin Y, Li J, Yang Y, Zhang M. Microplastics in three types of human arteries detected by pyrolysis-gas chromatography/mass spectrometry (Py-GC/MS). J Hazard Mater. 2024 May 5;469:133855. doi: 10.1016/j.jhazmat.2024.133855. Epub 2024 Feb 21. PMID 38428296
- [Background] Wang T, Yi Z, Liu X, Cai Y, Huang X, Fang J, Shen R, Lu W, Xiao Y, Zhuang W, Guo S. Multimodal detection and analysis of microplastics in human thrombi from multiple anatomically distinct sites. EBioMedicine. 2024 May;103:105118. doi: 10.1016/j.ebiom.2024.105118. Epub 2024 Apr 13. PMID 38614011
- [Background] Lee DH. Microplastics and Cardiovascular Diseases: Importance of Coexisting Environmental Pollutants. Circulation. 2024 Sep 17;150(12):908-910. doi: 10.1161/CIRCULATIONAHA.124.069801. Epub 2024 Sep 16. No abstract available. PMID 39283932
- [Background] Yang Y, Zhang F, Jiang Z, Du Z, Liu S, Zhang M, Jin Y, Qin Y, Yang X, Wang C, Gao H. Microplastics are associated with elevated atherosclerotic risk and increased vascular complexity in acute coronary syndrome patients. Part Fibre Toxicol. 2024 Aug 21;21(1):34. doi: 10.1186/s12989-024-00596-4. PMID 39164741
- [Background] Zhu X, Wang C, Duan X, Liang B, Genbo Xu E, Huang Z. Micro- and nanoplastics: A new cardiovascular risk factor? Environ Int. 2023 Jan;171:107662. doi: 10.1016/j.envint.2022.107662. Epub 2022 Nov 26. PMID 36473237
- [Background] Prattichizzo F, Ceriello A, Pellegrini V, La Grotta R, Graciotti L, Olivieri F, Paolisso P, D'Agostino B, Iovino P, Balestrieri ML, Rajagopalan S, Landrigan PJ, Marfella R, Paolisso G. Micro-nanoplastics and cardiovascular diseases: evidence and perspectives. Eur Heart J. 2024 Oct 7;45(38):4099-4110. doi: 10.1093/eurheartj/ehae552. PMID 39240674
- [Background] Marfella R, Prattichizzo F, Sardu C, Fulgenzi G, Graciotti L, Spadoni T, D'Onofrio N, Scisciola L, La Grotta R, Frige C, Pellegrini V, Municino M, Siniscalchi M, Spinetti F, Vigliotti G, Vecchione C, Carrizzo A, Accarino G, Squillante A, Spaziano G, Mirra D, Esposito R, Altieri S, Falco G, Fenti A, Galoppo S, Canzano S, Sasso FC, Matacchione G, Olivieri F, Ferraraccio F, Panarese I, Paolisso P, Barbato E, Lubritto C, Balestrieri ML, Mauro C, Caballero AE, Rajagopalan S, Ceriello A, D'Agostino B, Iovino P, Paolisso G. Microplastics and Nanoplastics in Atheromas and Cardiovascular Events. N Engl J Med. 2024 Mar 7;390(10):900-910. doi: 10.1056/NEJMoa2309822. PMID 38446676